CLINICAL TRIAL: NCT05906459
Title: Establishment of Rapid Diagnostic Procedure of "HCV Single-sample Detection Platform" in China
Brief Title: Simplification and Test and Treat Strategies Towards Hepatitis C Eliminationplatform" in China(STAT)
Acronym: STAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases Affiliation: Huashan Hospital, Huashan Hospital
Other Study IDs: STAT
Record Dates: First submitted 2023-05-29; First posted 2023-06-15 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C Virus Infection; Rapid diagnostic tests, RDTs; Anti-HCV antibody; HCV core antigen
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti-HCV antibody and HCV core antigen testing — HCV antibody screening were carried out with rapid diagnostic testings (RDTs) by colloidal gold method, using fingertip blood or residual blood from other testings.
  For samples with positive HCV antibody RDTs screening results, HCV core antigen detection will be carried out subsequently as diagnostic test. HCV core antigen detection will be conducted with chemiluminescent particle immunoassay using residual blood from other testings.

SUMMARY:
The present study aims to establish a " one-sample testing platform " and assess the prevalence of hepatitis C in individuals taking routine physical examination or outpatient visit in mainland China.

DETAILED DESCRIPTION:
Investigators intend to establish a one-sample testing platform to improve diagnosis and linkage to care process in participants under routine physical examination or outpatient visit. The platform is based on rapid diagnostic tests (RDTs) for HCV screening and HCV core antigen for confirmation. RDTs was used to screen for anti-HCV antibodies. The result of RDT will be interpreted within 15 minutes with the sensitivity of 98.9% (95%CI, 94.5% to 99.8%) and specificity of 98.9% (95%CI, 97.5% to 99.9%) using whole blood or finger-stick blood sample [3-5]. HCV core antigen is a marker of HCV replication and has a good correlation with HCV RNA in HCV-positive patients (R=0.98). A recent study suggested HCV core antigen testing could be used alternative testing for HCV RNA testing for diagnosis when HCV RNA testing was unavailable. The process of HCV core antigen test only takes 2-3 hours. "one-sample" means only one drop (10ul) of finger-stick blood or residual blood samples from other routine tests collected from patients was needed for anti-HCV antibody testing and HCV core antigen testing, which means they will not have to take another venepuncture. In addition, the use of RDT and HCV core antigen are also less costly. This approach might improve access to care, particularly in low-income and middle-income countries.

The present study aims to establish a " one-sample testing platform " in several medical institution to assess the prevalence of hepatitis C in individuals taking routine physical examination and further promote rapid diagnosis platform in mainland China, so as to achieve the goal in 2030.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years of age and older, regardless of age or gender.
* 2) The residual blood sample needs to be not less than 1ml.
* 3) Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* 1) Pregnant, lactating female and who is planning pregnancy during study period.
* 2) History of tumor or other severe, life-threating diseases.
* 3) Samples not meet collection requirements.
* 4) repeated enrollment.
* 5) HCV infection has been diagnosed.
* 6) Recent HCV RNA testing confirmed that there is no HCV infection.

Termination criteria:

* 1) Subject asked to withdraw consent.
* 2) Subjects may suffer adverse impact from the study at investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study plans to screen 20,000 subjects for anti-HCV from multiple centers across the country (including those who have physical examinations)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Completion rate of rapid diagnostic processes | 1day
  Completion rate of rapid diagnostic processes

SECONDARY OUTCOMES:
The prevalence of HCV infection | 1 day
  The prevalence of HCV infection in the population attending each center (including physical examination)
The proportion of abnormal fibroscan results, liver function, blood routine, and ultrasound data in HCV-infected people | 30 days
  For example, the confirmed rate of HCV infection in the screening population was much higher than that of HCV infection in the region in the epidemiological survey, and the degree of liver fibrosis and cirrhosis assessed by the confirmed population through this process was significantly lower than the mean HCV population reported in the literature, which indirectly reflected the potential benefit of rapid diagnosis process in helping to detect HCV infection missed in routine visits (including physical examination).
Additional time required by the testing process | 1 day
  Additional time required by the testing process
The feedback and evaluation from study participants | 1 day
  Feedback and assessments of study participants were collected using the Clinical Trial Participant Satisfaction Questionnaire (including whether it affects routine visits (including physical examination) procedures, and the acceptance of this process, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: WenHong Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (3):
- China (3):
  - The fifth People's Hospital Of Shanghai, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai, Shanghai, Shanghai Municipality
  - The First People's Hospital Of YunNan, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense the study will be published internationally to be available for the public.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within four year
Access Criteria: Not yet

REFERENCES:
- [Result] Shah H, Bilodeau M, Burak KW, Cooper C, Klein M, Ramji A, Smyth D, Feld JJ; Canadian Association for the Study of the Liver. The management of chronic hepatitis C: 2018 guideline update from the Canadian Association for the Study of the Liver. CMAJ. 2018 Jun 4;190(22):E677-E687. doi: 10.1503/cmaj.170453. No abstract available. PMID 29866893
- [Result] Mane A, Sacks J, Sharma S, Singh H, Tejada-Strop A, Kamili S, Kacholia K, Gautam R, Thakar M, Gupta RS, Gangakhedkar R. Evaluation of five rapid diagnostic tests for detection of antibodies to hepatitis C virus (HCV): A step towards scale-up of HCV screening efforts in India. PLoS One. 2019 Jan 17;14(1):e0210556. doi: 10.1371/journal.pone.0210556. eCollection 2019. PMID 30653562
- [Result] Chevaliez S, Roudot-Thoraval F, Hezode C, Pawlotsky JM, Njouom R. Performance of rapid diagnostic tests for HCV infection in serum or plasma. Future Microbiol. 2021 Jul;16:713-719. doi: 10.2217/fmb-2020-0295. Epub 2021 Jul 6. PMID 34227402
- [Result] Florea D, Neaga E, Nicolae I, Maxim D, Popa M, Otelea D. Clinical usefulness of HCV core antigen assay for the management of patients with chronic hepatitis C. J Gastrointestin Liver Dis. 2014 Dec;23(4):393-6. doi: 10.15403/jgld.2014.1121.234.chcv. PMID 25531997
- See also: Guidelines for the prevention and treatment of hepatitis C (2019 version) — http://www.lcgdbzz.org/custom/news/id/10075
- See also: Comparison between Colloidal Gold and Enzyme-linked Immunosorbent Assay of Hepatitis C Virus Antibody — https://gffhc975c3444c2dc4daasn9xfkk5n6p6v6xocfffi.res.gxlib.org.cn/periodical/ChlQZXJpb2RpY2FsQ0hJTmV3UzIwMjMwNDI2Eg95bGJqcWoyMDExMDUwMjkaCHg0aDN5Znoz